CLINICAL TRIAL: NCT05185999
Title: A Phase 1 Interventional Study to Test Short-Term Safety, Tolerability and Preliminary Efficacy of Sodium-Free Intraperitoneal 30% Icodextrin/10% Dextrose Solution in Peritoneal Dialysis Patients
Brief Title: Icodextrin Study to Test Short-Term Safety, Tolerability and Preliminary Efficacy of Sodium-Free Solution in PD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 119910
Record Dates: First submitted 2021-12-06; First posted 2022-01-11 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Failure
Keywords: Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Icodextrin; Glucose

STUDY DESIGN:
Intervention Model Description: Single-arm, Open Label, Phase 1 Interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intraperitoneal infusion with 500 mL of sodium-free 30% Icodextrin/ 10% Dextrose solution
  Interventions: Drug: Icodextrin/Dextrose

INTERVENTIONS:
Drug: Icodextrin/Dextrose — Single 8 hour dwell of a 500mL intraperitoneal sodium-free 30% Icodextrin / 10% Dextrose solution

SUMMARY:
Patients with kidney failure rely on dialysis for sodium and fluid removal. The importance of a sodium and fluid balance in patients with kidney disease is very important. Excess volume has been consistently associated with cardiovascular morbidity and mortality.

Many peritoneal dialysis (PD) patients need large volumes of dextrose or Icodextrin based solutions to achieve fluid removal. Commonly used PD solutions also have high sodium concentrations to limit sugar absorption. These PD fluids can reduce the amount of sodium removed and may eventually lead to water retention over time with possible adverse outcomes.

This research study is being conducted to determine if a single eight-hour dwell of intraperitoneal sodium-free 30% Icodextrin / 10% Dextrose solution is safe, tolerable and effective in achieving sodium and volume removal in PD patients.

DETAILED DESCRIPTION:
This study is a phase 1 interventional study in Peritoneal Dialysis Patients. Investigators will recruit 10 participants. This study involves one visit at the London Health Sciences Centre University Hospital lasting approximately 9 hours.

Study participants will receive one in-center PD dwell, consisting of peritoneal instillation of a sodium-free 30% Icodextrin/10% dextrose solution via their Tenckhoff catheter; the solution will be dwelling in the study participant's peritoneal cavity for a maximum of 8 hours as tolerated, at the end of which the solution will be drained.

Participants will be monitored during administration of the study solution, during dwell and up to one hour after the Peritoneal Dialysis fluid is drained.

Study participants will also undergo:

* Clinical blood pressure and heart rate monitoring: baseline + every 15 minutes for the first two hours; then every 30 minutes up until 1 hour post complete peritoneal solution drain
* Continuous Finapress hemodynamic monitoring (until 1 hour post peritoneal solution drain)
* Pain Monitoring throughout the study visit (Five point verbal scale and McGill Pain Questionnaire)
* Blood collection: baseline, 1, 2, 4, 8 hours into the dwell and 1 hour after the end of drain
* Peritoneal dialysate collection: 1, 2, 4, 8 hours into the dwell
* Urine collection throughout visit.

ELIGIBILITY:
Inclusion Criteria:

* Functioning Tenckhoff catheter
* Stable PD prescription regimen (continuous ambulatory PD or automated PD) for the past month
* Age 18 years or older
* Willing and able to provide informed consent
* Able to Speak and Read English

Exclusion Criteria:

* Type 1 or uncontrolled diabetes mellitus
* Active infections
* Pre-study serum sodium <130 mmol/L
* Serum bicarbonate < 18mmol/L
* Patients with standard PD prescriptions relying exclusively on lowest glucose containing fluid
* Allergy to starch-based polymers (e.g. corn starch) and/or icodextrin
* Intolerance to maltose or isomaltose
* Glycogen storage disease
* Uncorrectable mechanical defects that prevent effective PD or increase the risk of infection
* Documented loss of peritoneal function or extensive adhesions that compromise peritoneal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related Adverse Events or Serious Adverse Events. | Throughout the study visit - approximately 9 hours
  Adverse Events and Serious Adverse Events will help determine the safety of the intraperitoneal solution. Change in symptoms from baseline.
Changes in hemodynamic stability (Blood Pressure) | Throughout the study visit - approximately 9 hours
  This will determine participant tolerability of the treatment. Systolic and Diastolic blood pressure (mm/Hg) will be measured throughout the study visit at baseline, every 15 minutes for 2 hours, then every 30 minutes until 1 hour after solution drain is complete.
  If the systolic or diastolic blood pressure changes more then 40 mmHg or more at any time point the study physician will be consulted for direction.
Changes in hemodynamic stability (Heart Rate) | Throughout the study visit - approximately 9 hours
  This will determine participant tolerability of the treatment. We will monitor heart rate (bpm) at baseline, every 15 minutes for 2 hours, then every 30 minutes until 1 hour after solution drain is complete.
  If heart rate is less then 50 beats per minute or greater then 120 beats per minute the study physician will be alerted.
Changes in hemodynamic stability (Finapres monitoring) | Throughout the study visit - approximately 9 hours
  This will determine tolerability of the treatment. Hemodynamic monitoring using Finapres (finger-cuff to detect beat-to-beat changes) Hemodynamic variables such as pulse rate, blood pressure, stroke volume, cardiac output, and total peripheral resistance are derived. (for post hoc observational analysis only)
Sodium Removal | Throughout the study visit - approximately 9 hours
  This will measure the efficacy of the treatment. Serum sodium (mmol/L) levels will be drawn at baseline, 1, 2, 4, 8 and 9 hours and sent to the lab for analysis.
Pain Assessment (Five-point Verbal Scale) | Throughout the study visit - approximately 9 hours
  This pain assessment will determine tolerability of the treatment. Five-point Verbal Scale (0-no pain, 1=mild pain, 2=moderate pain, 3=severe pain, 4=very severe pain)
  We will complete the Five-point Verbal Scale at the following time points:
  * start of infusion at 1, 3, and 5 minutes after start of infusion and at end of infusion of the Icodextrin/Dextrose solution
  * 15, 30 minutes into dwell, hourly during dwell and at the end of dwell of the Icodextrin/Dextrose solution
  * start of drain, 5 minutes into drain and end of drain of the Icodextrin/Dextrose solution If Five-Point verbal scale >3 for two consecutive readings and if pain exceeds individual tolerability, fluid will be drained and the study physician will be alerted.
Pain Assessment (McGill Pain Questionnaire) | Throughout the study visit - approximately 9 hours
  This pain assessment will determine tolerability of the treatment. McGill Pain Questionnaire (MPQ) 30 minutes into dwell of the Icodextrin/Dextrose solution The MPQ explores the multi-dimensional nature of pain.
Ultrafiltration Volume | Throughout the study visit - approximately 9 hours
  This will measure the efficacy of the treatment. Ultrafiltrate will be measured in litres post drain.

SECONDARY OUTCOMES:
Serum Glucose monitoring and glucose absorption | Throughout the study visit - approximately 9 hours
  This will measure glucose (mmol/L) levels will be drawn at baseline, 1, 2, 4, 8 and 9 hours and sent to the lab for analysis.
Dialysate icodextrin biproducts | Throughout the study visit - approximately 9 hours
  This will measure the efficacy of the treatment. A 15 ml sample of peritoneal effluent will be collected at 1, 2, 4 and 8 hours in to dwell. This sample will be sent to the lab for the analysis of dialysate Icodextrin biproducts.
Serum Icodextrin biproducts | Throughout the study visit - approximately 9 hours
  This will measure the efficacy of the treatment. Serum will be collected at baseline, 1, 2, 4 and 8 and 9 hours and sent to lab for analysis of Icodextrin biproducts.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, MD/PHD, Principal Investigator — London Health Sciences Centre - Victoria Hospital
Locations (2):
- Canada (2):
  - Victoria Hospital, London Health Sciences Centre, London, Ontario
  - Westmount Kidney Care Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No